CLINICAL TRIAL: NCT02029118
Title: Effect of Acupoint Application With Herbal Medicine in Patients With Stable Angina Pectoris: Randomized, Controlled,Double Blind Clinical Study
Brief Title: Acupoint Application in Patients With Stable Angina Pectoris (AASAP)
Acronym: AASAP
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Chengdu University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2011SZ0302.2
Record Dates: First submitted 2013-11-24; First posted 2014-01-07 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Stable Angina Pectoris
Keywords: Acupoint Application,Stable Angina Pectoris,herbal medicine
MeSH Terms: conditions — Angina, Stable | interventions — storax; isoborneol; Frankincense; Leeching; Acupuncture Points; Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Herbal application on acupoint group (Experimental): Containing the herbal medicine application on the specific acupoints plus foundation treatment
  Interventions: Drug: Herbal plaster ( styrax, borneol, frankincense, santalum,trichosanthes kirilowii Maxim, allium macrostemon Bunge, leech); Device: acupoint; Drug: Aspirin: 100mg qd; Metoprolol：25mg bid; Ramipril:5mg qd; Atorvastatin:20mg qn.
- Placebo application on acupoint (Placebo Comparator): Not containing herbal medicine application on the specific acupoints plus foundation treatment
  Interventions: Device: acupoint; Drug: Aspirin: 100mg qd; Metoprolol：25mg bid; Ramipril:5mg qd; Atorvastatin:20mg qn.
- Herbal application on non-acupoint group (Placebo Comparator): Containing the herbal medicine application on the non-acupoints plus foundation treatment
  Interventions: Drug: Herbal plaster ( styrax, borneol, frankincense, santalum,trichosanthes kirilowii Maxim, allium macrostemon Bunge, leech); Drug: Aspirin: 100mg qd; Metoprolol：25mg bid; Ramipril:5mg qd; Atorvastatin:20mg qn.
- Placebo application on non-acupoint (Sham Comparator): Not containing herbal medicine application on the non-acupoints plus foundation treatment
  Interventions: Drug: Aspirin: 100mg qd; Metoprolol：25mg bid; Ramipril:5mg qd; Atorvastatin:20mg qn.

INTERVENTIONS:
Drug: Herbal plaster ( styrax, borneol, frankincense, santalum,trichosanthes kirilowii Maxim, allium macrostemon Bunge, leech) — Application containing herbal medicine that mainly include styrax, borneol, frankincense, santalum,trichosanthes kirilowii Maxim, allium macrostemon Bunge, leech and other herbal medicine.
  Other Names: Herbal medicine application
  Arms: Herbal application on acupoint group; Herbal application on non-acupoint group
Device: acupoint — select acupoint according to traditional Chinese medicine
  Other Names: acupuncture point
  Arms: Herbal application on acupoint group; Placebo application on acupoint
Drug: Aspirin: 100mg qd; Metoprolol：25mg bid; Ramipril:5mg qd; Atorvastatin:20mg qn. — foundation treatment
  Other Names: basic treatment

SUMMARY:
Hypothesis: acupoint application is effective for managing chronic stable angina pectoris. Aim: to evaluate the efficacy and safety of acupoint application on the specific acupoints for chronic stable angina pectoris. Design: A Randomized, Controlled,Double Blind trial. 200 participants will be included. Four arms: herbal medicine application on acupoint group , placebo application on acupoint group , herbal medicine application on non-acupoint group and placebo application on non-acupoint group.

DETAILED DESCRIPTION:
Acupoint application with herbal medicine is a kind of external treatment of traditional Chinese medicine and has a long history in China, which is use herbal medicine made of plaster and stick to specific acupoints, using the double effects of acupoints and herb to treat disease. In China, acupoint application with herbal medicine has been used in clinical treatment of angina pectoris, but there is no convincing evidence for the efficacy of acupoint application for angina pectoris, due to low methodologic quality and small sample size. The investigators designed the Randomized, Controlled, Double Blind clinical trial to investigates the efficacy of acupoint application in treating angina pectoris, the purpose of this study is to provide the convincing evidence for acupoint application treatment of angina pectoris.

ELIGIBILITY:
Inclusion Criteria:

1.Meet the diagnostic criteria of American College of Cardiology(ACC)/American Heart Association (AHA) angina pectoris of coronary heart disease.

2.35 ≤ age ≤ 85 years, both male and female.

3.The onset of angina pectoris≥3 months, and the frequency of angina attack≥2 a week.

4.Patients signed the informed consent

Exclusion Criteria:

1. age≤35 or age≥85.
2. Pregnant women or women in lactation or women of child bearing potential plan to conceive in the recent six months.
3. history of diabetes.
4. Co-infection or bleeding, allergic.
5. Currently participating in other clinical trials

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2012-10; Primary Completion 2015-05 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Number of angina attacks at 12 weeks | at baseline,4, 8weeks after inclusion
  The change frequency of angina attack during every 4-week.

SECONDARY OUTCOMES:
Change from Baseline the severity of angina ( VAS score) at 12 weeks | at baseline,4, 8weeks after inclusion
  The VAS score evaluation angina pain severity
Change from Baseline the dosage of nitroglycerin at 12 weeks | at baseline,4, 8weeks after inclusion
  Observed reduction in the dose of nitroglycerin
Seattle Angina Questionnaire | at baseline,4, 8weeks after inclusion
self-rating anxiety scale | at baseline,4, 8weeks after inclusion
Self-rating Depression Scale | at baseline,4, 8weeks after inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Fanrong Liang, Principal Investigator — Chengdu University of TCM
Locations (1):
- Affiliated hospital of Chengdu University of TCM, Chengdu, Sichuan, China

REFERENCES:
- [Derived] Li DH, Xie J, Ren YL, Zheng H, Lyu JL, Leng JY, Zhang LL, Zhang J, Fan HL, Liang FR. Effectiveness and Safety of Acupoint Application of Guan Xin Su He Pill () for Patients with Chronic Stable Angina Pectoris: A Multi-Center, Randomized Controlled Trial. Chin J Integr Med. 2021 Nov;27(11):838-845. doi: 10.1007/s11655-021-2870-3. Epub 2021 Aug 13. PMID 34387828
- [Derived] Ren Y, Li D, Zheng H, Lv J, Leng J, Zhang L, Zhang J, Fan H, Liang F. Acupoint application in patients with chronic stable angina pectoris: study protocol of a randomized, double-blind, controlled trial. Evid Based Complement Alternat Med. 2014;2014:619706. doi: 10.1155/2014/619706. Epub 2014 Aug 27. PMID 25250055